CLINICAL TRIAL: NCT06339775
Title: Blinatumomab Sequential Donor Lymphocyte Infusion in Acute B Lymphocytic Leukemia Observation of Therapeutic Effect in Patients With Recurrence After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Blinatumomab for Relapsed Acute B Lymphoblastic Leukemia After Transplantation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Suping ZHANG (Other)
Responsible Party: Sponsor-Investigator, Suping ZHANG, visiting staff, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024318
Record Dates: First submitted 2024-03-18; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Acute B-cell Lymphoblastic Leukemia
Keywords: Acute B-cell lymphoblastic leukemia; Relapse; allogeneic hematopoietic stem cell transplantation; Blinatumomab
MeSH Terms: conditions — Recurrence | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab followed by donor lymphocyte infusion (Experimental): Patients with positive MRD were treated with Blinatumomab 28μg×5-15 days, followed by DLI treatment.
  (MNC infusion is about 5×10^7/kg~1×10^8/kg). Patients with hematologic recurrence were given Blinatumomab 9μg D1-4,11.66μg d5-7,28μg Starting from d8 （8 to 21 days in total）, followed by DLI treatment (infusion of MNC approximately 5×10^7/kg~1×10^8/kg).
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — patients with positive MRD were treated with Blinatumomab 28μg×5-15 days, followed by DLI treatment.
  (MNC infusion is about 5×10^7/kg~1×10^8/kg). Patients with hematologic recurrence were given Blinatumomab 9μg D1-4,11.66μg d5-7,28μg Starting from d8 （8 to 21 days in total）, followed by DLI treatment (infusion of MNC approximately 5×10^7/kg~1×10^8/kg).
  Other Names: donor lymphocyte infusion

SUMMARY:
B-ALL patients received regular follow-up after allogeneic hematopoietic stem cell transplantation, and in case of recurrence, they were given Blinatumomab.

Anti-treatment was followed by DLI, and the second course was performed 1-2 months after DLI.

Patients with positive MRD were treated with Blinatumomab 28μg×5-15 days, followed by DLI treatment.

(MNC infusion is about 5×10^7/kg~1×10^8/kg). Patients with hematologic recurrence were given Blinatumomab 9μg D1-4,11.66μg d5-7,28μg Starting from d8 （8 to 21 days in total）, followed by DLI treatment (infusion of MNC approximately 5×10^7/kg~1×10^8/kg). Objective To observe and analyze the efficacy and side effects of Blinatumomab followed by donor lymphocyte infusion in patients with relapsed acute B lymphoblastic leukemia after allogeneic hematopoietic stem cell transplantation in our hospital.

DETAILED DESCRIPTION:
Patients with acute B-cell lymphoblastic leukemia who relapsed after receiving allogeneic hematopoietic stem cell transplantation in our hospital and received sequential donor lymphocyte infusion （DLI） treatment after relapse. The patients with acute B-cell lymphoblastic leukemia who relapsed after receiving allogeneic hematopoietic stem cell transplantation in our hospital from September 2023 to December 2026 and received sequential donor lymphocyte infusion （DLI） treatment after relapse were enrolled.

1. Age ≤65 years old
2. Stable vital signs
3. No severe infection
4. No grade II-IV graft-versus-host disease
5. No organ failure

Exclusion criteria

1. Age >65 years old
2. Unstable vital signs
3. Complicated with severe infection
4. Complicated with grade II-IV graft-versus-host disease
5. Organ failure such as heart, liver, kidney, etc.
6. Complicated with central nervous system leukemia
7. Drug allergy to the treatment regimen Treatment regimen B-ALL patients were regularly followed up after allogeneic hematopoietic stem cell transplantation. When relapse occurred, Blinatumomab was given sequentially after DLI, and the second course of treatment was conducted 1-2 months after DLI.

MRD-positive patients were given Blinatumomab 28μg×5-15 days, followed by DLI treatment （infusion of MNC is about 5×10^7/kg~1×10^8/kg）.

Hematologic relapse patients were given Blinatumomab 9μg d1-4,11.66μg d5-7,28μg d8 （a total of 8 to 21 days）, followed by DLI treatment （infusion of MNC is about 5×10^7/kg~1×10^8/kg）. The duration of using Blinatumomab was determined according to the patient's tolerance, economic situation and other comprehensive factors.

Main observation and statistical indicators Overall survival after relapse, disease-free survival, incidence of cytokine release syndrome （CRS）, incidence of acute/chronic graft-versus-host disease （GVHD） after treatment, incidence of infection, incidence of hematological adverse reactions, etc.Compared with patients receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤65 years old
2. Stable vital signs
3. No severe infection
4. There was no grade II-IV graft-versus-host disease
5. No organ failure

Exclusion Criteria:

1. Age > 65 years old
2. Unstable vital signs
3. Complicated with severe infection
4. Combined with grade Ⅱ-Ⅳ graft-versus-host disease
5. Heart, liver, kidney and other organ failure
6. Complicated with central nervous system leukemia
7. Allergies to medications in the treatment regimen

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | three years
  Survival time of patients with recurrence after treatment
Disease-free survival | three years
  Disease-free survival time after treatment for relapsed patients

SECONDARY OUTCOMES:
incidence of cytokine release syndrome （CRS） | 2 weeks later
  Recurrent patients received treatment 2 weeks later
Incidence of acute/chronic graft-versus-host disease （GVHD） | 2 weeks later
  Recurrent patients received treatment 100 days later.
hematological adverse reactions Incidence rate | 2 weeks later
  Recurrent patients received treatment 2 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Zhilei BIAN, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhenzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT06339775/Prot_000.pdf
  • Informed Consent Form (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT06339775/ICF_001.pdf